# 受试者知情同意书

项目名称: 一项多中心内镜下内痔微创治疗复发率的回顾性研究

方案版本号及版本日期: V2.0/2023-11-14

知情同意书版本号及版本日期: V2.0/2023-11-14

## 尊敬的受试者:

我们邀请您参加一项研究,该本研究已经得到南方医科大学深圳医院医学伦理委员会的审查和批准。在您作决定之前,我们希望您能了解开展本研究的原因以及它需要您做的事情。您参加本研究纯属自愿,也就是说您既可以选择参加,也可以选择不参加。研究团队将会为您讲解本信息告知书,并解答您的任何疑问。

如果您有任何不清楚的地方,请向我们提问。欢迎您与伴侣、家人、朋友和医生等与您关系亲近的人讨论本研究及本文件所含的信息。

在您考虑了与本研究相关的所有信息,并且您的所有问题都得到解答后,如果您同意参加,则在进行任何研究相关的程序之前,研究团队会请您签署知情同意书并注明日期(在本文件末尾)。

## 一、研究背景

本研究的研究背景是内镜下内痔微创治疗术在全国各级医院积极推广,本项目负责人获得 2021 年度广东省卫生健康适宜推广项目(20216252151077306),随着项目的推广,我们发现该技术的安全性、有效性及中长期的复发率尚缺乏大宗数据的研究,因此,我们对本中心 3 年来开展的内镜下内痔微创治疗病例资料进行梳理,回顾性分析此项技术的应用情况,希望借此探讨内痔微创治疗复发的相关因素,依据复发率与时间的关系等多因素,为内痔微创治疗术后随访的时间及序贯治疗的方案提供可参考数据。

内痔是直肠下端黏膜下齿状线上方及肛门皮肤处的静脉丛充血、静脉曲张而形成的柔软静脉丛。目前已证实,内镜下内痔微创治疗对 I-III 度有症状的内痔是有效且安全的。I-III 度内痔合并便血以硬化剂注射治疗为主,II、III 期内痔合并脱垂以套扎治疗为主。内镜下硬化剂注射治疗是指内镜辅助下向粘膜下层注射

硬化剂,使痔核缩小。内镜下套扎术是指用套扎器将直肠肛管粘膜套扎起来,使 其直肠壁纤维化,不仅可以防止脱垂,还可以减少血液流入痔疮静脉丛,达到止 血的目的。

目前内镜下内痔微创治疗术开展时间尚短,其长期有效率及复发率是一个备受关注的问题,一些医患对此技术的疗效存在质疑。为此,笔者查阅大量文献,发现关于该技术复发率的数据鲜有报道,特别是引起内镜下内痔微创治疗复发的相关因素亦无研究,这给临床医生开展工作带来极大不便,在与患者制定手术方案过程中强调新技术的应用,而未告知存在复发的风险以及可能需要二次手术的干预,致使患者未享受合理知情权,满意度降低,医患双方获益不大。结合上述情况考量,本研究着眼于术后疗效与复发率的数据分析,试图寻找内镜下内痔微创治疗术的复发因素。

#### 二、研究目的

本研究的研究目的是

主要目的:观察各种内镜下内痔微创治疗方式以及不同时间点的内镜下内痔 微创治疗对 I 度-III 度内痔患者的短期、长期复发率

次要目的: 观察内镜下内痔微创治疗术的安全性和有效性

#### 三、研究产品(或诊疗技术)介绍

本研究是针对 I-III 度内痔、存在内镜下内痔微创治疗指征的患者,进行硬化剂注射治疗(采取聚桂醇原液,于痔核基底部口侧及肛侧 1-6 个位点注射,观察痔核实变情况,必要时术中补充治疗)、套扎治疗(利用七环套扎器于痔上粘膜及痔核多点套扎,观察痔核回纳情况)、套扎联合硬化剂注射治疗(利用七环套扎器于痔上粘膜及痔核多点套扎,观察痔核回纳情况,如仍有红色征则补充硬化剂注射治疗)。

### 四、研究过程

#### 1.多少人将参与这项研究?

大约超过615人会在本院参与本研究。

### 2.研究步骤

### ■研究开始前

为检查您是否适合参加,本次筛选将进行以下程序:

- 获取您的人口统计学特征和生命体征
- •对您进行体格检查,主要包括肛门视诊及直肠指诊
- •询问您的病史相关信息和伴随用药
- •采集血液进行实验室检测
- ●如果您是有生育可能的女性,将进行妊娠检测。您的妊娠检测结果必须为 阴性才能参加本研究。

筛选的检查结果和/或相关问题的结果将帮助研究人员决定您是否可以继续本研究。如果这些检查表明您适合参加本研究,研究人员将通知您尽快进行访视 2。如果您不满足相关标准,则不能继续参与本次研究,研究人员也会第一时间 将结果通知到您。

### ■基线期

如果研究人员确认您符合加入本试验,您则确定被纳入本研究根据不同的内 镜下内痔微创治疗的方式记录。本次访视将进行以下程序:

- •再次确认您是否具备参加本次研究的资格
- •分配给您参加本次研究特定的识别号
- •根据微创治疗方式记录组别
- •进行体格检查并采集生命体征数据

#### ■治疗期

•对您进行体格检查并采集生命体征数据

#### ■随访期

您完成该阶段的访视以后,通常认为您已经完成了整个研究,研究人员将在 此期间执行以下程序:

术后1天、7天及1个月、小于6个月、6至12个月以及12个月以上接受 微信问卷调查、电话等方式对您进行随访,内容包括术后出血、疼痛、脱垂、 排尿评分,判断有无血栓性外痔情况。

#### 3、本研究会进行哪些检测和评估?

在提供书面知情同意后,本研究期间您将进行一些检测、检查和程序。如果 您对其中的任何检测有任何疑虑,请和研究医生讨论。

关于本研究的检测和程序, 我们想对您做如下说明:

• 病史: 研究医生会询问您一些问题, 了解任何当前或既往疾病, 以及用药

史、手术史、月经史等。

- 人口统计资料:研究医生将收集有关您个人的信息,如出生日期和族裔背景。
- 体检: 研究医生将对您的身体进行医学检验来评估下列全部或部分人体系统: 头部、眼睛、耳鼻喉、胸、肺、心脏、腹部、骨骼、皮肤、颈部、肛门和神经系统。
  - 身高和体重: 将测量您的身高和体重。
  - 生命体征: 研究医生将测量您的血压、心率、体温和呼吸率。
- 抽血:本研究期间仅在术前一次抽血(如果术后有感染迹象,发热等,则需要复测化验)。将为下列项目采集血液样本:

血常规、凝血四项、感染八项。

- 尿液常规检查。
- 调查问卷。

## 3.这项研究会持续多久?

本次临床研究共约 12 个月以上(6 次访视),分为 1 次手术治疗与 1 个月跟踪访视。在加入本研究期间,您必须配合术后 1 天、7 天及 1 个月、小于 6 个月、6 至 12 个月以及 12 个月以上接受访视。

您可以在任何时间选择退出研究而不受到任何惩罚,也不会丧失您本应获得的任何利益。然而,如果在研究途中您决定退出本研究,我们鼓励您先和您的医生商议。考虑到您的安全性问题,有可能在退出后,会进行一次相关检查。

### 五、风险和/或不适

研究团队的主要目标是始终保证您的安全。然而,内镜下内痔微创治疗后随 访可能会引起副作用,包括罕见或目前未知的副作用。在本研究期间,我们将利 用验血和验尿、体检来密切监测您的各项指标,以及其它身体系统。

如果您感觉您的健康状况有任何恶化,或者您出现意外或异常的症状,应立即联系研究团队,即使您认为这些问题并非由研究程序造成。

研究程序带来的风险和不适,如:

5.1 血液采集: 血液样本将通过插入您的手臂或手部静脉内的小针头采集。

在插入和拔出针头时您可能会感到不适和/或酸痛,并有可能出现小的瘀伤。在 极少数情况下,静脉可能堵塞,或者可能发生小的神经损伤,导致麻木和疼痛。 如果发生这种情况,一段时间后会消退。

5.2 微信或电话随访:可能随访时耽误您的私人时间,干扰到您的情绪。我们会将随访流程简介,减少您的不良情绪发生,并安抚您的情绪。

## 六、参加研究有什么受益?

参加本临床试验的受试者预期有直接获益,可能的获益如下:有助于了解内镜下内痔微创治疗获益情况,有利于了解该治疗方式复发率,有利于此种治疗的复发时间,并精致采取复发前于预性治疗。

本临床试验可能的间接受益,您的参与有助于推动内镜下内痔微创治疗的方法学革新,进而协助临床医生降低医疗费用,具有极其重要的现实意义。我们希望从您参与的本研究中得到的信息有助于将来为该疾病的患者开发出新疗法。

## 七、备选的治疗方案

除了参与本研究,您有如下选择方案:不采用此随访研究方案,患者可自行来门诊就诊随访。

您可随时与研究医生讨论您的疾病及其可能引起的结果,并确定选取哪一种作为您的最佳治疗方案。

# 八、研究结果的使用和个人信息的保密

在研究结束时,我们会撰写一份报告并发送给政府监管机构。本研究的结果也可能在期刊上发表,可能在会议上报告,但不会包含任何可能识别您身份的信息。

为保证隐私,出于研究目的发布的记录或样本不会附上您的姓名及其它身份识别信息。相反,您的信息将仅通过一个代码标识。只有研究医生和授权人员能够通过一份清单把此代码与您的姓名联系起来,该清单将在研究中心安全地保存。

可能为了确保研究是否在研究中心正确进行,必要时申办者、伦理审查委员

会以及政府管理部门按规定可以查阅您的资料,他们受保密义务约束,不会侵犯您的隐私。

您有权控制对您个人信息的使用和披露。在国家法律允许的情况下,您可以 随时要求查看您的医疗信息。您有权通过研究医生查看所收集的有关您的所有信 息,并要求进行纠正(如果适用)。

# 九、研究相关新信息

研究期间,若有研究程序变化、新发现的副作用或可能影响您健康或参加意愿的重大情况出现,研究小组将通知您。研究医生会立即通知您,还会与您一起讨论您是否想继续参加本研究。如果您决定不再继续参加本研究,研究医生会做出安排,让您的诊疗护理继续下去。如果您决定留在本研究中,研究医生可能会要求您签署一份新的知情同意书。

## 十、关于研究费用、补偿以及损害赔偿

### 1. 研究所用的药物及相关检查费用

本临床试验的费用全部由受试者自行承担(包括术前常规化验检查、肠镜检查、 麻醉费、内镜下微创治疗手术费、耗材费等)。

#### 2. 参加研究的补偿

参加本研究您不会得到任何经济补偿

### 3. 损害赔偿

若因为临床试验造成了意外伤害,我们会提供必要的医疗措施(如采血化验,在插入和拔出针头时您可能会感到不适和/或酸痛,并有可能出现小的瘀伤,本研究中心负责处理伤口等),并根据我国相关法规条例规定,承担相应的医疗费用及对此提供相应的经济补偿。

### 十一、受试者的权利和责任

#### 1. 您的权利

在参加研究的整个过程中,您都是自愿的。如果您决定不参加本研究,也不会影响您应该得到的其他治疗。如果您决定参加,会要求您在这份书面知情同意书上签字。您有权在试验的任何阶段随时退出试验而不会遭到歧视或受到不公平的待遇,您相应医疗待遇与权益不受影响。

## 2. 您的责任

需要提供有关自身病史和当前身体状况的真实情况;告诉研究医生自己在本次研究期间所发现的任何不适;在任何的实验性治疗中都有可能对您或您的胎儿造成风险,所以,您和您的伴侣在研究期间均应避免任何可能会导致怀孕的活动。若是您在研究过程中怀孕,请立即通知您的研究医生。

## 十二、相关联系方式

如果您有与本研究相关的任何问题,请通过微信/电话 <u>13384662039</u> 与<u>朱颖</u>联系。

如果您有与自身权利/权益相关的任何问题,或者您想反映参与本研究过程中遭遇的困难、不满和忧虑,或者想提供与本研究有关的意见和建议,请联系南方医科大学深圳医院医学伦理委员会,联系电话: 0755-23360060, 电子邮箱: szyyec@163.com

# 受试者签字页

# 知情同意声明

我已被告知此项研究的目的、背景、过程、风险及获益等情况。我有足够的 时间和机会进行提问,问题的答复我很满意。

我也被告知, 当我有问题、想反映困难、顾虑、对研究的建议, 或想进一步 获得信息,或为研究提供帮助时,应当与谁联系。

我知道我可以选择不参加此项研究,或在研究期间的任何时候无需任何理由 退出本研究。此外,研究者没有对我使用欺骗、利诱、胁迫等手段强行让我同意 参加研究。

我已知道如果我的状况更差了,或者我出现严重的不良反应,或者我的研究 医生觉得继续参加研究不符合我的最佳利益,他/她会决定让我退出研究。无需 征得我的同意,资助方或者监管机构也可能在研究期间终止研究。如果发生该情 况, 医生将及时通知我, 研究医生也会与我讨论我的其他选择。

我已经阅读这份知情同意书,并且同意参加本研究。

我将得到这份知情同意书的副本,上面包含我和研究者的签名。

| 受试者签名:<br>联系电话: | 日期: |
|------------------|----------------------|
| <b>状</b> 尔·巴伯: | |
| 法定代理人签字: | 日期: |
| 联系电话: | |
| (注:如果受试者无行为能力或限制 | 引行为能力时,如纳入精神障碍/意识不清等 |
| 弱势群体则需法定代理人在以下法定 | (代理人签字处签名) |
| 公平见证人签名: | 日期: |
| 联系电话: | |
| (注:仅当可能纳入有知情能力,但 | 无法阅读文本的受试者(如:文盲、视力障 |
| 碍)时,才需要公平见证人签名,见 | 证人知情时研究者最好留取视频材料作为知 |
| 情证据)。 | |
| 我已准确地将这份文件告知受证 | 【者,他/她准确地阅读了这份知情同意书, |
| 并证明该受试者有机会提出问题,他 | 」/她是自愿同意的。 |
| 研究者签名: | _ 日期: |
| 联系电话: | |